CLINICAL TRIAL: NCT04834375
Title: Randomized Open Investigation Determining Steroid Dose (ROIDS-Dose)
Brief Title: Randomized Open Investigation Determining Steroid Dose
Acronym: ROIDS-Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Stella S Hahn, MD, Associate Medical Director, Northwell Sleep Disorders Center, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0171
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Covid19
Keywords: dexamethasone; COVID-19; COVID pneumonia; respiratory failure; steroids
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a parallel fashion into either the standard dexamethasone dose of 6 mg or weight-based dexamethasone of 0.2 mg/kg (maximum dose of 20 mg)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard dexamethasone dose (No Intervention): Dexamethasone 6 mg IV daily for 10 days
- Weight-based dexamethasone dose (Experimental): Dexamethasone 0.2 mg/kg/day IV (maximum 20 mg daily) for 10 days
  Interventions: Drug: Weight-based dexamethasone dose

INTERVENTIONS:
Drug: Weight-based dexamethasone dose — Weight-based dexamethasone dose in COVID-19 patients with hypoxic respiratory failure
  Other Names: Higher dexamethasone dose
  Arms: Weight-based dexamethasone dose

SUMMARY:
Dexamethasone has been approved for the treatment of severe COVID-19, but higher doses of steroids may be more effective. The purpose of this research study is to compare the current standard dose of dexamethasone 6 mg to a higher, weight-based dosing (0.2 mg/kg with maximum dose of 20 mg) to determine if it would be more effective against COVID-19 pneumonia.

DETAILED DESCRIPTION:
Treatment for COVID-19 patients with respiratory failure has been vexing, but the use of steroids has shown promise. In a recent randomized control trial, dexamethasone 6 mg once daily showed a modest decrease in mortality among hospitalized COVID-19 patients who require oxygen supplementation or invasive mechanical ventilation. Other trials have shown that the inflammatory response to COVID-19 can be further attenuated at higher dosages of dexamethasone. These higher dosages have not been well studied and have not been directly compared to the current standard dose of dexamethasone 6 mg daily. We propose that a higher dexamethasone dose, equivalent to methylprednisolone 1 mg/kg/day which is routinely used to treat other inflammatory conditions of the lungs, may be more effective than the current standard dose in reducing mortality in COVID-19 patients with respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater or equal than 18 years old
* COVID-19 infection confirmed by positive PCR test
* Hypoxemia defined by an oxygen saturation < 94% or the need for supplemental oxygen

Exclusion Criteria:

* Corticosteroid use for > 48h within the past 15 days prior to enrollment
* Use of steroids with doses higher than the equivalent to dexamethasone 6 mg
* Use of immunosuppressive drugs
* Pregnant women
* Chronic oxygen use
* Known history of dexamethasone allergy
* DNR / DNI
* Patient or proxy cannot consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mangala Narasimhan, DO, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] WHO Rapid Evidence Appraisal for COVID-19 Therapies (REACT) Working Group; Sterne JAC, Murthy S, Diaz JV, Slutsky AS, Villar J, Angus DC, Annane D, Azevedo LCP, Berwanger O, Cavalcanti AB, Dequin PF, Du B, Emberson J, Fisher D, Giraudeau B, Gordon AC, Granholm A, Green C, Haynes R, Heming N, Higgins JPT, Horby P, Juni P, Landray MJ, Le Gouge A, Leclerc M, Lim WS, Machado FR, McArthur C, Meziani F, Moller MH, Perner A, Petersen MW, Savovic J, Tomazini B, Veiga VC, Webb S, Marshall JC. Association Between Administration of Systemic Corticosteroids and Mortality Among Critically Ill Patients With COVID-19: A Meta-analysis. JAMA. 2020 Oct 6;324(13):1330-1341. doi: 10.1001/jama.2020.17023. PMID 32876694
- [Background] Tomazini BM, Maia IS, Cavalcanti AB, Berwanger O, Rosa RG, Veiga VC, Avezum A, Lopes RD, Bueno FR, Silva MVAO, Baldassare FP, Costa ELV, Moura RAB, Honorato MO, Costa AN, Damiani LP, Lisboa T, Kawano-Dourado L, Zampieri FG, Olivato GB, Righy C, Amendola CP, Roepke RML, Freitas DHM, Forte DN, Freitas FGR, Fernandes CCF, Melro LMG, Junior GFS, Morais DC, Zung S, Machado FR, Azevedo LCP; COALITION COVID-19 Brazil III Investigators. Effect of Dexamethasone on Days Alive and Ventilator-Free in Patients With Moderate or Severe Acute Respiratory Distress Syndrome and COVID-19: The CoDEX Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1307-1316. doi: 10.1001/jama.2020.17021. PMID 32876695
- [Background] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Background] Edalatifard M, Akhtari M, Salehi M, Naderi Z, Jamshidi A, Mostafaei S, Najafizadeh SR, Farhadi E, Jalili N, Esfahani M, Rahimi B, Kazemzadeh H, Mahmoodi Aliabadi M, Ghazanfari T, Sattarian M, Ebrahimi Louyeh H, Raeeskarami SR, Jamalimoghadamsiahkali S, Khajavirad N, Mahmoudi M, Rostamian A. Intravenous methylprednisolone pulse as a treatment for hospitalised severe COVID-19 patients: results from a randomised controlled clinical trial. Eur Respir J. 2020 Dec 24;56(6):2002808. doi: 10.1183/13993003.02808-2020. Print 2020 Dec. PMID 32943404
- [Derived] Rabascall CX, Lou BX, Dhar S, Hasan Z, Fryman C, Izard S, Makaryus M, Acharya S, Mastroianni F, Kamper M, Duenas S, Gong J, Shah D, Khanijo S, Ying D, Habibullah J, Kim DH, Butzko R, Oks M, Birnbaum B, Moore J, Singh AK, Quintero L, Lau M, Honigman J, Hilewitz A, Shah K, Simonson J, Agrawal A, Frank M, Tsegaye A, Narasimhan M, Greenberg H, Hahn SS. Randomized Open Investigation Determining Steroid Dose in Severe COVID-19: The ROIDS-Dose Clinical Trial. Cureus. 2022 Nov 4;14(11):e31086. doi: 10.7759/cureus.31086. eCollection 2022 Nov. PMID 36475114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients underwent screening and randomization between March 19, 2021 and December 28, 2021 at seven hospitals in Northwell Health in New York. Randomization was performed using a computer-generated allocation sequence via the Research Electronic Data Capture (REDCap) system. Eligible patients were randomized in a 1:1 ratio stratified by the trial site to either the standard dose group or the intervention group.
Period: Overall Study
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Started | 72 | 70
Completed | 72 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.22 (15.18) | 55.46 (15.11) | 56.35 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 49 | 50 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 56 | 55 | 111
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 26 | 51
  White | 27 | 25 | 52
  More than one race | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Steroid initiation prior to the study [Count of Participants; unit: Participants] | 68 | 66 | 134
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.72 (8.99) | 33.57 (9.84) | 32.62 (9.43)
Dexamethasone dose [Mean (Standard Deviation); unit: mg] | 6 (0) | 17.49 (2.66) | 11.66 (6.06)
Pre-enrollment nadir oxygen saturation [Mean (Standard Deviation); unit: % of oxygen saturation] | 83.92 (10.72) | 84.43 (7.96) | 84.17 (9.43)
Oxygen required on enrollment [Count of Participants; unit: Participants] | 72 | 70 | 142
Oxygen modality on enrollment [Count of Participants; unit: Participants]
  Nasal cannula | 42 | 49 | 91
  Venturi mask | 1 | 1 | 2
  Non-rebreather mask | 9 | 5 | 14
  High flow nasal cannula | 14 | 11 | 25
  Non-invasive ventilation | 2 | 3 | 5
  Mechanical ventilation | 4 | 1 | 5
Charlson comorbidity index [Mean (Standard Deviation); unit: units on a scale] — Scale used to predict 10-year survival in patients with multiple comorbidities. Ranges from a minimum of 0 points to a maximum of 37 points. The higher the score, the worse estimated 10-year survival.
  units on a scale | 2.18 (1.92) | 1.90 (1.95) | 2.04 (1.93)
4C mortality score [Mean (Standard Deviation); unit: units on a scale] — Score used to predict in-hospital mortality in patients admitted with COVID-19. Ranges from a minimum of 0 points to a maximum of 21 points.
  0-3 points: Low risk (1.2 - 1.7% in-hospital mortality) 4-8 points: Intermediate risk (9.1 - 9.9% in-hospital mortality) 9-14 points: High risk (31.4 - 31.9% in-hospital mortality) 15-21 points: Very high risk (61.5% - 66.2% in-hospital mortality)
  units on a scale | 8.67 (3.69) | 7.86 (3.52) | 8.27 (3.62)
Other treatments for COVID-19 [Count of Participants; unit: Participants]
  Tocilizumab | 18 | 17 | 35
  Remdesivir | 65 | 65 | 130
  Monoclonal antibodies | 0 | 2 | 2
  Any COVID-19 vaccination | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality at 28 Days
Description: All cause mortality at 28 days.
  Comment: Primary outcome was all cause mortality at 28 days but the patients were followed until end of admission for the final disposition (death or discharge) which accounts for the differences in the primary outcome of mortality at 28 days and the total number of deaths at discharge
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 15 | 12

2. Secondary Outcome: Number of Participants Admitted to the ICU
Description: Number of participants that required admission to the ICU
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 27 | 12

3. Secondary Outcome: Days of Stay in the Intensive Care Unit
Description: ICU length of stay
Time Frame: 28 days
Population: Among patients admitted to the ICU
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 27 | 12
days | 15.33 (11.28) | 11.33 (8.85)

4. Secondary Outcome: Days of Hospitalization
Description: Duration of hospitalization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
days | 14.83 (17) | 11.56 (8.88)

5. Secondary Outcome: Number of Participants That Required Higher Levels of Oxygen Supplementation
Description: Venturi mask, Non-rebreather mask, High-flow nasal cannula, Non-invasive ventilation
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 32 | 31

6. Secondary Outcome: Number of Participants That Required Invasive Mechanical Ventilation
Description: Escalation to invasive mechanical ventilation
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 19 | 10

7. Secondary Outcome: Duration of Invasive Mechanical Ventilation
Description: Total days requiring invasive mechanical ventilation
Time Frame: 28 days
Population: Among patients requiring invasive mechanical ventilation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 23 | 11
days | 19.95 (16.14) | 10.90 (8.88)

8. Secondary Outcome: Number of Participants That Required ECMO
Description: Refractory hypoxemia requiring ECMO
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 3 | 2

9. Secondary Outcome: Number of Participants That Required Tracheostomy
Description: Need for tracheostomy
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 5 | 1

10. Secondary Outcome: Number of Participants That Developed Secondary Bacterial or Fungal Infections
Description: Culture positive evidence of secondary bacterial or fungal infections
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 19 | 9

11. Secondary Outcome: Number of Participants That Developed Clinically Significant Hyperglycemia
Description: Defined as need for insulin drip or ICU admission to control hyperglycemia
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants | 5 | 4

12. Secondary Outcome: Number of Participants That Required Oxygen Supplementation a Discharge From the Hospital
Description: Need for oxygen supplementation at hospital discharge
  Comment: Corrected total number of discharged patients alive to 55 in the "Standard Dexamethasone Dose" Arm.
Time Frame: Until hospital discharge
Population: Among patients discharged alive
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 55 | 58
Participants | 25 | 27

13. Secondary Outcome: Subjective Symptoms at 28 Days
Description: Subjective symptoms questionnaire at 28 days
Time Frame: 28 days
Population: Among patients alive at 28 days with a completed response
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 36 | 46
Participants
  Better | 33 | 44
  Same/worse | 3 | 2

14. Secondary Outcome: Disposition Upon Discharge
Description: Home, home with physical therapy, other (skilled nursing facility, long-term acute care facility, long-term care facility / nursing home, acute rehabilitation facility, hospice care), expired
Time Frame: At hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
Number analyzed (Participants) | 72 | 70
Participants
  Home | 40 | 42
  Home with physical therapy | 10 | 11
  Other | 5 | 5
  Expired | 17 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 28 days. Mortality was assessed through 28 days for the primary outcome but final disposition was assessed at end of hospitalization (e.g. death or discharge).
Arm/Group | Standard Dexamethasone Dose | Weight-based Dexamethasone Dose
All-Cause Mortality (participants affected / at risk) | 17/72 | 12/70
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/70
Other Adverse Events (participants affected / at risk) | 24/72 | 13/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dexamethasone Dose (N=72) | Weight-based Dexamethasone Dose (N=70)
Clinically significant hyperglycemia (Endocrine disorders) | 5 | 4 — Development of clinically significant hyperglycemia, defined as requiring ICU admission for treatment of hyperglycemia or requirement of an insulin infusion
Secondary bacterial or fungal infections (Infections and infestations) | 19 | 9

LIMITATIONS AND CAVEATS:
Study was not blinded. Small sample size may have reduced the ability to detect statistically significant differences among some of the secondary outcomes. Selecting a maximum dose of 20 mg in the weight-based dexamethasone group may have affected the results. As the standard of care for the treatment of COVID-19 changed over time, those changes may have affected patient care in undetectable ways, affecting the results of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04834375/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04834375/ICF_001.pdf